CLINICAL TRIAL: NCT04758442
Title: Optimal Dosing of Vancomycin in an Adult Population of Hemato-oncology: a Nomogram Based on a Bayesian Population Model to Predict Initial Dosage of Vancomycin
Brief Title: Optimal Dosing of Vancomycin in an Adult Population of Hemato-oncology
Acronym: Hemato-Vanco
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-2482
Record Dates: First submitted 2021-02-09; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Vancomycin; Hematologic Malignancies; Febrile Neutropenia
Keywords: Bayesian model; Pharmacokinetics
MeSH Terms: conditions — Hematologic Neoplasms; Febrile Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vancomycin (Experimental): Subjects with hematologic cancer who received intravenous vancomycin for a suspected or confirmed infection.
  Interventions: Other: Additional blood sample

INTERVENTIONS:
Other: Additional blood sample — Included subjects will provided three blood samples to follow vancomycin concentration

SUMMARY:
This is a single-center prospective pharmacokinetic study. The principal objective is to collect new data among patients with hematologic cancer to develop a Bayesian population pharmacokinetic model and to improve dose adjustment of intravenous vancomycin. Approximately 40 subjects meeting the inclusion and no exclusion criteria will be enrolled in the study. Vancomycin blood concentration will be measured at steady-state at three different moment for each participant : immediately before the infusion, 1 hour after the infusion and during the elimination phase (at 3, 4 or 5 hours after the infusion). This additional vancomycin serum concentration in the elimination phase will be used to estimate more precisely the vancomycin pharmacokinetic parameters in this specific population including the distribution volume and the elimination of the molecule. Ultimately, the purpose of this study is to create a nomogram to predict the optimal initial vancomycin dosing in adult patients with a hematologic cancer.

DETAILED DESCRIPTION:
STUDY DESIGN:

Prospective, monocentric, pharmacokinetic study.

Adults who have been diagnosed with a hematologic malignancy, are hospitalized at Maisonneuve-Rosemont hospital and received at least 3 doses of intravenous vancomycin.

Pharmacokinetic parameters: Serum vancomycin concentration measured at steady state just before the beginning of the infusion (trough), 1 hour after completion of the infusion (peak) and between 3 to 5 hours after the end of the infusion (additional blood draw during the elimination phase).

RECRUITMENT PROCESS:

A systematic daily screening of hospitalized patients diagnosed with a hematologic cancer will be made by the research team and the pharmacists 7 days a week. An information sheet will be given to all potential eligible patients at their admission. When intravenous vancomycin is prescribed, a member of the research team will explain the study and present the Information and Consent Form (ICF) to the potential participant to obtain his/her official informed consent.

DATA COLLECTION:

Three blood draws will be planned around the fourth or fifth dose of vancomycin and collected by the nursing team. The sampling scheme is as follows: just before the beginning of the infusion (trough), 1 hour after completion of the infusion (peak) and 3, 4 or 5 hours after the end of the infusion (additional blood draw during the elimination phase) according to the assigned time of the participant. The assigned time of the additional blood draw will be randomized at the inclusion of the subject in the study. A member of the research team will provide the tubes to the nurse, will write and save sampling times and will ship the blood samples to the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 and over;
* Subjects diagnosed with a hematologic cancer;
* Subjects hospitalized at Maisonneuve-Rosemont hospital between February 2021 and August 2021;
* Intravenous vancomycin treatment prescribed by a doctor;
* Subjects received at least 3 doses of intravenous vancomycin.

Exclusion Criteria:

* Non-malignant diagnosis (aplastic anemia and rare metabolic diseases);
* Subjects admitted to a critical care unit;
* End-stage renal disease (GFR < 15 mL/min/1.73m2);
* Patients undergoing dialysis/renal replacement therapy;
* Acute kidney injury at the moment of the first vancomycin dosage (definition adapted from KDIGO criteria):

  1. Increase in serum creatinine by ≥ 26.5 umol/L within 48 hours or
  2. Increase in serum creatinine to ≥ 1.5 times baseline within prior 7 days
* Pregnant women;
* Severely burn patients;
* Inability to give free and informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic Parameters : Volume of Distribution | During intravenous vancomycin treatment assessed to 72 hours
  Estimated from vancomycin serum concentrations and patient characteristics
Pharmacokinetic Parameters : Vancomycin clearance | During intravenous vancomycin treatment assessed to 72 hours
  Estimated from vancomycin serum concentrations and patient characteristics

SECONDARY OUTCOMES:
Area Under the concentration-time Curve (AUC) | between 0 to 24 hours during vancomycin administration
Serum Vancomycin Through Concentration | 5 minutes before the selected infusion
  Vancomycin concentration measured just before the next infusion
Serum Vancomycin Peak Concentration | 60 minutes after the end of the infusion
  Vancomycin concentration measured 1 hour after the end of vancomycin infusion
Serum Vancomycin Elimination Phase Concentration | 3 to 5 hours after the end of the infusion (+/- 30 minutes)
  Vancomycin concentration measured 3 to 5 hours after the end of vancomycin infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Freifeld AG, Bow EJ, Sepkowitz KA, Boeckh MJ, Ito JI, Mullen CA, Raad II, Rolston KV, Young JA, Wingard JR; Infectious Diseases Society of America. Clinical practice guideline for the use of antimicrobial agents in neutropenic patients with cancer: 2010 update by the infectious diseases society of america. Clin Infect Dis. 2011 Feb 15;52(4):e56-93. doi: 10.1093/cid/cir073. PMID 21258094
- [Background] Wingard JR, Hsu J, Hiemenz JW. Hematopoietic stem cell transplantation: an overview of infection risks and epidemiology. Infect Dis Clin North Am. 2010 Jun;24(2):257-72. doi: 10.1016/j.idc.2010.01.010. PMID 20466269
- [Background] Rybak M, Lomaestro B, Rotschafer JC, Moellering R Jr, Craig W, Billeter M, Dalovisio JR, Levine DP. Therapeutic monitoring of vancomycin in adult patients: a consensus review of the American Society of Health-System Pharmacists, the Infectious Diseases Society of America, and the Society of Infectious Diseases Pharmacists. Am J Health Syst Pharm. 2009 Jan 1;66(1):82-98. doi: 10.2146/ajhp080434. No abstract available. PMID 19106348
- [Background] Pfizer Canada Inc. PRODUCT MONOGRAPH : VANCOMYCIN HYDROCHLORIDE FOR INJECTION, USP. Kirkland, QC Pfizer Canada Inc.;2018.
- [Background] Rybak MJ. The pharmacokinetic and pharmacodynamic properties of vancomycin. Clin Infect Dis. 2006 Jan 1;42 Suppl 1:S35-9. doi: 10.1086/491712. PMID 16323118
- [Background] Zhao W, Zhang D, Fakhoury M, Fahd M, Duquesne F, Storme T, Baruchel A, Jacqz-Aigrain E. Population pharmacokinetics and dosing optimization of vancomycin in children with malignant hematological disease. Antimicrob Agents Chemother. 2014 Jun;58(6):3191-9. doi: 10.1128/AAC.02564-13. Epub 2014 Mar 24. PMID 24663023
- [Background] Okada A, Kariya M, Irie K, Okada Y, Hiramoto N, Hashimoto H, Kajioka R, Maruyama C, Kasai H, Hamori M, Nishimura A, Shibata N, Fukushima K, Sugioka N. Population Pharmacokinetics of Vancomycin in Patients Undergoing Allogeneic Hematopoietic Stem-Cell Transplantation. J Clin Pharmacol. 2018 Sep;58(9):1140-1149. doi: 10.1002/jcph.1106. Epub 2018 May 15. PMID 29762865
- [Background] Aljutayli A, Marsot A, Nekka F. An Update on Population Pharmacokinetic Analyses of Vancomycin, Part I: In Adults. Clin Pharmacokinet. 2020 Jun;59(6):671-698. doi: 10.1007/s40262-020-00866-2. PMID 32020531
- [Background] Marsot A, Boulamery A, Bruguerolle B, Simon N. Vancomycin: a review of population pharmacokinetic analyses. Clin Pharmacokinet. 2012 Jan 1;51(1):1-13. doi: 10.2165/11596390-000000000-00000. PMID 22149255
- [Background] Neely MN, Youn G, Jones B, Jelliffe RW, Drusano GL, Rodvold KA, Lodise TP. Are vancomycin trough concentrations adequate for optimal dosing? Antimicrob Agents Chemother. 2014;58(1):309-16. doi: 10.1128/AAC.01653-13. Epub 2013 Oct 28. PMID 24165176
- [Background] Bury D, Ter Heine R, van de Garde EMW, Nijziel MR, Grouls RJ, Deenen MJ. The effect of neutropenia on the clinical pharmacokinetics of vancomycin in adults. Eur J Clin Pharmacol. 2019 Jul;75(7):921-928. doi: 10.1007/s00228-019-02657-6. Epub 2019 Mar 15. PMID 30877327
- [Background] Jarkowski A 3rd, Forrest A, Sweeney RP, Tan W, Segal BH, Almyroudis N, Wang ES, Wetzler M. Characterization of vancomycin pharmacokinetics in the adult acute myeloid leukemia population. J Oncol Pharm Pract. 2012 Mar;18(1):91-6. doi: 10.1177/1078155211402107. Epub 2011 Apr 26. PMID 21521799
- [Background] Buelga DS, del Mar Fernandez de Gatta M, Herrera EV, Dominguez-Gil A, Garcia MJ. Population pharmacokinetic analysis of vancomycin in patients with hematological malignancies. Antimicrob Agents Chemother. 2005 Dec;49(12):4934-41. doi: 10.1128/AAC.49.12.4934-4941.2005. PMID 16304155
- [Background] Choi MH, Choe YH, Lee SG, Jeong SH, Kim JH. Neutropenia is independently associated with sub-therapeutic serum concentration of vancomycin. Clin Chim Acta. 2017 Feb;465:106-111. doi: 10.1016/j.cca.2016.12.021. Epub 2016 Dec 23. PMID 28025029
- [Background] Bosso JA, Nappi J, Rudisill C, Wellein M, Bookstaver PB, Swindler J, Mauldin PD. Relationship between vancomycin trough concentrations and nephrotoxicity: a prospective multicenter trial. Antimicrob Agents Chemother. 2011 Dec;55(12):5475-9. doi: 10.1128/AAC.00168-11. Epub 2011 Sep 26. PMID 21947388
- [Background] Taghizadeh-Ghehi M, Rezaee S, Gholami K, Hadjibabaie M. Predictive performance of Vancomycin population pharmacokinetic models in Iranian patients underwent hematopoietic stem cell transplantation. J Res Pharm Pract. 2015 Jul-Sep;4(3):129-34. doi: 10.4103/2279-042X.162357. PMID 26311080
- [Background] Monteiro JF, Hahn SR, Goncalves J, Fresco P. Vancomycin therapeutic drug monitoring and population pharmacokinetic models in special patient subpopulations. Pharmacol Res Perspect. 2018 Jul;6(4):e00420. doi: 10.1002/prp2.420. PMID 30156005